CLINICAL TRIAL: NCT00682994
Title: Patient and Family Decision Making and Information Disclosure Preferences in the Palliative Care Setting: a Multi-Center Survey in Chile, Guatemala, and U.S.
Brief Title: Patient and Family Decision Making in the Palliative Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2007-0667
Record Dates: First submitted 2008-05-15; First posted 2008-05-23 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2012-08

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Family Member; Palliative Care; Decision Making; Information Disclosure; Interview; Survey; Questionnaire
MeSH Terms: interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decision Making (Other): Questionnaire + Interview
  Interventions: Behavioral: Interview; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Interview — Interview lasting about 5-10 minutes.
Behavioral: Questionnaire — Questionnaires taking 20-30 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this research study is to learn about any differences in certain health-related preferences between patients with cancer and their families.

The main preferences being studied are how decisions are made about healthcare, as well as how much information people want to know about cancer.

Specifically, researchers will compare questionnaire and interview data from Hispanic-Americans living in the United States (the M. D. Anderson part of this multicenter study) with Hispanics living in Latin America (in particular, Argentina, Chile, and Guatemala).

DETAILED DESCRIPTION:
Study Background:

People from different cultures may have different preferences in the way decisions about their healthcare are made, as well as how much information they may want to know about the diseases they may have. However, patients and families sometimes disagree about these preferences. In this study, researchers want to learn about any differences in healthcare decision-making and information-sharing preferences between patients and their families, among a group of people from different Hispanic backgrounds.

(Please note that the phrase "family member" has been used in this consent form for short, but the definition includes non-family members that you may consider a "significant other").

Screening Procedures:

Participants in this study must also agree to give the name of a family member (a parent, spouse, adult child, sibling, other family member, or a non-family member that you consider a "significant other") that researchers can ask to participate in a separate part of this study that will require signing a separate consent form. (If the person of your choice is not with you at the time of joining the study, he/she may come back to the clinic at your next follow-up visit.)

If the family member agrees, he/she will complete a similar series of questionnaires about his/her preferences in decisions about your healthcare, what information he/she might want you to know about the disease, and what information he/she might want to know about the disease him/herself. Like you, he/she will also be asked how decisions about your healthcare have been made, his/her satisfaction with those decisions and your healthcare, and his/her sense of connection with what he/she defines to be the overall Hispanic culture. He/she will also complete a similar interview on general information (such as marital status and educational level).

Study Visit:

If you agree to take part in this study and you have given the name of a family member, you will be interviewed to ask for general information about yourself ("demographic" information such as marital status and educational level).

After that, you will complete a series of questionnaires that ask about your preferences in decisions about your healthcare and what information you may want to know about the disease, how decisions about your healthcare have been made, your satisfaction with those decisions and your healthcare, and your sense of connection with what you define to be the overall Hispanic culture.

It should take about 5-10 minutes for the interview and another 20-30 minutes to complete the questionnaires.

Your interview and questionnaire responses will not be shared with your regular doctor. If you feel you need a doctor's opinion about anything that is asked about in the interview and/or questionnaires, please contact your doctor.

Family Member's Participation:

Your family member would complete the questionnaires separately and be interviewed separately from you. You may ask as many additional family members as needed, until one agrees. However, if the family member is scheduled for his/her study visit but does not end up completing the study procedures (interview and questionnaires), your interview and questionnaire data will be destroyed without being used in this study.

Confidentiality:

Your interview and questionnaire responses will only be used for this research study, and will not be shared with your family member.

Length of Study Participation:

After completing the interview and questionnaires, your participation in this study will be over.

This is an investigational study. In total, up to 900 patients and family members will take part in this multicenter study. Up to 300 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with advanced cancer (local recurrence or metastatic) at the time of their follow up visit to the outpatient palliative care clinic or at an agreed date after the first visit to the outpatient palliative care clinic.
2. Patient designates a family member who is a patient's parent, spouse, adult child, sibling, other relative, or significant other (any other person defined by the patient as a partner) to answer the family questionnaire.
3. Patient is 18 years of age or older (as the assessment tools used in this study have not been validated in the pediatric population).
4. Patient with normal cognitive status as determined by the interviewer and by her/his ability to understand the nature of the study and consent process.
5. Patient willing to participate in the study and sign informed consent.
6. Family member is 18 years of age or older (as the assessment tools used in this study have not been validated in the pediatric population).
7. Family member with normal cognitive status as determined by the interviewer and by her/his ability to understand the nature of the study and consent process.
8. Family member willing to participate in the study and sign informed consent.
9. All participants in the international centers must be from Argentinian, Chilean, or Guatemalan descendence respectively.
10. All participants in the U.S. must be from self-reported Hispanic descendence, first or second generation immigrants, and reside in the U.S. for at least 5 years.

Exclusion Criteria:

1. Either patient or family member can not complete the assessments independently.
2. Either patient or family member refuses to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2008-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Differences in Proportions of Preference for Passive Decision Making | 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- UT MD Anderson Cancer Center, Houston, Texas, United States
- Fundacion FEMEBA - Programa Argentino de Medicina Paliativa - Hospital Tornu, Buenos Aires, Argentina
- Dr. Sotero del Rio Hospital - Catholic University of Chile, Santiago, Chile
- Guatemalan Cancer Institute - INCAN, Guatemala City, Guatemala

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org